CLINICAL TRIAL: NCT02892461
Title: Effect of Umbilical Cord Milking on Iron Related Health Outcomes for Cesarean-Delivered Infants: A Randomized Controlled Trial
Brief Title: Effect of Umbilical Cord Milking on Iron Related Health Outcomes for Cesarean-Delivered Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Hunan Provincial Maternal and Child Health Care Hospital (Other); Liuyang Maternal and Child Health Care Hospital (Unknown)
Responsible Party: Principal Investigator, Jianmeng Liu, Professor in Epidemiology and Biostatistics; Director of Institute of Reproductive and Child Health, Peking University; Director of Office for National Maternal and Child Health Statistics of China, Peking University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 81571517
Record Dates: First submitted 2016-08-23; First posted 2016-09-08 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Anemia, Iron-Deficiency
Keywords: Anemia, Iron-Deficiency; Cesarean Section; Umbilical Cord Milking; Randomized Controlled Trial
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Umbilical cord milking (Experimental): The cord will be cut at 25 cm from the umbilical stump within 30 seconds after the infant is taken out from the uterus and its blood will be milked to the infant gently and thoroughly in 30 seconds during resuscitation on the radiant warmer, and then the cord will be cut at 2 to 3 cm from the umbilical stump.
  Interventions: Procedure: Umbilical cord milking
- Routine clinical treatment and care (No Intervention): The cord will be dealt with routine clinical method, which means it will be cut twice within 1minute after the infant is taken out from the uterus, the first cut is on the operating table, while the second cut is on the radiant warmer.

INTERVENTIONS:
Procedure: Umbilical cord milking — As same as that in arm descriptions.
  Arms: Umbilical cord milking

SUMMARY:
This study aims to determine whether umbilical cord milking can improve iron related health outcomes for cesarean-delivered infants. Half of participants will receive umbilical cord milking, while the other half will receive routine clinical treatment and care.

DETAILED DESCRIPTION:
In recent years, several professional organizations have recommended delayed cord clamping to improve placental transfusion for newborns born vaginally based on a series of randomized controlled studies. However, no similar recommendations are available for cesarean-delivered infants. Investigators found that cesarean-delivered infants were more vulnerable to iron deficiency and anemia compared with those born vaginally, suggesting that it is urgently needed to find a similar anemia prevention strategy for infants born by cesarean sections.

In this study, investigators aim to test whether umbilical cord milking (UCM), a potentially promising strategy for cesarean delivery, can improve iron related health outcomes for cesarean-delivered infants. A total of 450 term pregnant women who are planning to give births by cesarean sections will be enrolled from two hospitals in Hunan province and randomly assigned to either UCM group or control group. Infants will be followed up at 1, 6, 12, 18 months for the evaluation of the impact of UCM on iron deficiency, anemia, as well as growth and the developmental status of language and mental/behavioral outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Full-term pregnancy (no less than 37 gestational weeks)
* Cesarean section before the labor starts or cesarean section after the labor starts but with cervix less than 3 cm
* Plan to take vaccines and receive routine child health care in the hospital where she gives birth

Exclusion Criteria:

* Maternal hypertensive disorder
* Gestational diabetes with macrosomia
* Gestational diabetes with polyhydramnios
* Maternal severe anemia with hemoglobin less than 70 g/L
* Maternal coagulation disorders
* Fetal growth restriction
* Major congenital anomalies
* Hemolytic disease of the newborn or hydrops fetalis
* Short umbilical cord length (< 30 cm)
* Severe cord or placenta abnormalities such as cord prolapse, true knots, placental abruption and placenta previa
* Other conditions that are not suitable for the study judged by the doctors

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 484 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Change in infant's serum ferritin (μg/L) | At birth (baseline), 6 and 12 months after birth
  At birth (baseline)-2 ml umbilical cord blood, 6 and 12 months old-2 ml infant's venous blood for each measure.

SECONDARY OUTCOMES:
Change in infant's erythrocyte counts (10^12/L) | At birth (baseline), 1, 6 and 12 months after birth
  At birth (baseline)-1 ml umbilical cord blood, 1 month old-20 μL infant's peripheral blood of finger, 6 and 12 months old-1 ml infants' venous blood for each measure.
Change in infant's hemoglobin concentration (g/L) | At birth (baseline), 1, 6 and 12 months after birth
  A participant's erythrocyte counts and hemoglobin concentration are detected using the same blood sample.
Change in infant's hematocrit (%) | At birth (baseline), 1, 6 and 12 months after birth
  A participant's erythrocyte counts, hemoglobin concentration and hematocrit are detected using the same blood sample.
Change in infant's weight (kg) | At birth (baseline), 1, 6, 12 and 18 months after birth
  Every infant's weight will be measured twice each time, but if the difference between the two measurement results is more than 0.1 kg, it will be measured for the third time.
Change in infant's height (cm) | At birth (baseline), 1, 6, 12 and 18 months after birth
  Every infant's height will be measured twice each time, but if the difference between the two measurement results is more than 0.5 cm, it will be measured for the third time.
Infant's language development | 18 months old
  The infant's development status of language will be assessed by the Language Developmental Survey (LDS).
Infant's mental/behavioral development | 18 months old
  The infant's mental/behavioral development will be assessed by the Child Behavior Checklist (CBCL).
Change in infant's transcutaneous bilirubin concentration (mg/dL) | 1 (baseline), 2, 3, 4 and 5 days after birth
  An infant's transcutaneous bilirubin concentration will be detected for five days after birth with time recorded. To ensure accuracy, each time it will be repeatedly detected for three times.
Number of infants with neonatal jaundice in the experimental group and the control group | Up to 18 months old
  At each follow-up visit (1, 6, 12 and 18 months after birth), parents will be asked whether their children suffer from jaundice up to then. If so, the doctor will ask them about the onset time, possible causes, treatment and prognosis of the disease.
Number of infants with polycythemia in the experimental group and the control group | Up to 18 months old
  At each follow-up visit (1, 6, 12 and 18 months after birth), parents will be asked whether their children suffer from polycythemia up to then.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmeng Liu, PhD, Study Chair — Peking University; Hongtian Li, PhD, Principal Investigator — Peking University; Yubo Zhou, PhD, Principal Investigator — Peking University; Qiyun Du, MD, Principal Investigator — Hunan Provincial Maternal and Child Health Care Hospital; Shujin Zhou, B.S.Med, Principal Investigator — Liuyang Maternal and Child Health Care Hospital
Locations (2):
- China (2):
  - Hunan Provincial Maternal and Child Health Care Hospital, Changsha, Hunan
  - Liuyang Maternal and Child Health Care Hospital, Guankou, Hunan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li HT, Trasande L, Zhu LP, Ye RW, Zhou YB, Liu JM. Association of cesarean delivery with anemia in infants and children in 2 large longitudinal Chinese birth cohorts. Am J Clin Nutr. 2015 Mar;101(3):523-9. doi: 10.3945/ajcn.114.092585. Epub 2014 Dec 24. PMID 25733637
- [Background] McDonald SJ, Middleton P, Dowswell T, Morris PS. Effect of timing of umbilical cord clamping of term infants on maternal and neonatal outcomes. Cochrane Database Syst Rev. 2013 Jul 11;2013(7):CD004074. doi: 10.1002/14651858.CD004074.pub3. PMID 23843134
- [Background] Hutton EK, Hassan ES. Late vs early clamping of the umbilical cord in full-term neonates: systematic review and meta-analysis of controlled trials. JAMA. 2007 Mar 21;297(11):1241-52. doi: 10.1001/jama.297.11.1241. PMID 17374818
- [Background] Perlman JM, Wyllie J, Kattwinkel J, Atkins DL, Chameides L, Goldsmith JP, Guinsburg R, Hazinski MF, Morley C, Richmond S, Simon WM, Singhal N, Szyld E, Tamura M, Velaphi S; Neonatal Resuscitation Chapter Collaborators. Part 11: Neonatal resuscitation: 2010 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. Circulation. 2010 Oct 19;122(16 Suppl 2):S516-38. doi: 10.1161/CIRCULATIONAHA.110.971127. No abstract available. PMID 20956259
- [Background] Committee on Obstetric Practice, American College of Obstetricians and Gynecologists. Committee Opinion No.543: Timing of umbilical cord clamping after birth. Obstet Gynecol. 2012 Dec;120(6):1522-6. doi: 10.1097/01.AOG.0000423817.47165.48. PMID 23168790
- [Background] McCAUSLAND AM, HOLMES F, SCHUMANN WR. Management of cord and placental blood and its effect upon the newborn. Calif Med. 1949 Sep;71(3):190-6. PMID 18137215
- [Background] SIDDALL RS, CRISSEY RR, KNAPP WL. Effect on cesarean section babies of stripping or milking of the umbilical cords. Am J Obstet Gynecol. 1952 May;63(5):1059-64. doi: 10.1016/0002-9378(52)90546-2. No abstract available. PMID 14923706
- [Background] Daniel DG, Weerakkody AN. Neonatal prevention of iron deficiency. Blood can be transfused from cord clamped at placental end. BMJ. 1996 Apr 27;312(7038):1102-3. doi: 10.1136/bmj.312.7038.1102d. No abstract available. PMID 8616446
- [Background] Upadhyay A, Gothwal S, Parihar R, Garg A, Gupta A, Chawla D, Gulati IK. Effect of umbilical cord milking in term and near term infants: randomized control trial. Am J Obstet Gynecol. 2013 Feb;208(2):120.e1-6. doi: 10.1016/j.ajog.2012.10.884. Epub 2012 Oct 31. PMID 23123382
- [Background] Mercer JS, Erickson-Owens DA. Rethinking placental transfusion and cord clamping issues. J Perinat Neonatal Nurs. 2012 Jul-Sep;26(3):202-17; quiz 218-9. doi: 10.1097/JPN.0b013e31825d2d9a. PMID 22843002